CLINICAL TRIAL: NCT04309708
Title: A Prospective, Randomized, Cntrolled, Multi-center Clinical Study on Efficacy and Safety of Infusion Therapy by Comparing Original Perfusor Line (Orange,Art No.8723017) With Original Perfusor Line (Black,Art No.8723010) in Pump Infusion.
Brief Title: Efficacy and Safety Assessment for a New UV-protected Pump Infusion Line in Intravenous Infusion Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Medical International Trading Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HC-G-H-1722
Record Dates: First submitted 2019-12-23; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Subarachnoid Hemorrhage
Keywords: pump infusion; photodegradation; IV infusion therapy
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: Randomized, Controlled, Parallel, Multi-center study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Original Perfusor Line(Art.No.8723017) (Experimental)
  Interventions: Device: Nimodipine pump infusion
- Original Perfusor Line(Art.No.8723010) (Active Comparator)
  Interventions: Device: Nimodipine pump infusion

INTERVENTIONS:
Device: Nimodipine pump infusion — Patients with nimodipine pump infusion with pump infusion line and other infusion equipments

SUMMARY:
To verify the efficacy and safety of Original Perfusor Line (Art.No.8723017) in infusion therapy in Patients with light sensitive drug infusion.

Subjects who choose to use Original Perfusor Line for their planned infusion treatment (nimodipine injection) as per the study protocol will be enrolled. The 300 subjects will be 1:1 randomized into the experimental group or the control group, using Original Perfusor Line (Art.No. 8723017) connected with an injection pump for infusion treatment with nimodipine injection or Original Perfusor Line (Art.No.8723010) connected with an injection pump for infusion treatment with nimodipine injection, respectively.Use of both the test product and the control product will be in strict accordance with their package insert.

The primary endpoint is the percentage of products which successful infuse fluids or medications into patient's circulatory system without leakage of fluids or medications, visible catheter embolism, air embolism and micro embolism in the infusion system and the secondary endpoint is the quality assessment for the clinical application of the products,such as the percentage of products which are qualified for infusion administration including link and removal, transparence, and tenacity.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years, all genders;
* Patients who will be treated plan to use injection pump for infusion treatment with nimodipine injection by infusion pump.
* Participated in this study voluntarily and signed informed consent form.

Exclusion Criteria:

* Patients have contraindication on Nimodipine.
* Patients allergic to polyethylene (PE) material;
* Patients with aspartate transaminase(AST) and alanine transaminase(ALT) are 2 times higher than normal range, Serum creatinine(Scr) is 1.5 times higher than normal range.
* Patient with malignant tumor, pregnant or Lactation;
* Patients had participated in other clinical trials within 1 month and in parallel with other trials;
* Patients are unsuitable to participate in this study as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-08 (Actual)

PRIMARY OUTCOMES:
Infusion success rate | 2 hours after infusion therapy completion
  The percentage of products which successful infuse fluids or medications into patient's circulatory system without leakage of fluids or medications

SECONDARY OUTCOMES:
Product pass rate | 2 hours after infusion therapy completion
  percentage of the quantity of products that pass the evaluation in the sum of products that pass the evaluation and products that fail the evaluation.

OTHER OUTCOMES:
Incidence of Adverse Events/Serious Adverse Events during treatment | Day -7 (At least 7days before infusion therapy) , Day 0 (infusion therapy), 2 hours after infusion therapy completion
Blood coagulation Test | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  Including tests of prothrombin time(PT) in second, activated partial thrombophastin time(APTT) in second and thrombin time(TT) in second
white blood cell(WBC) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in 10^9/L
Neutrophil(NEU) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in 10^9/L
Red blood cell(RBC) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in 10^12/L
Hemoglobin(HGB) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in g/L
Hematocrit(HCT) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in percentage(%)
Platelet(PLT) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in 10^9/L
Blood urea nitrogen(BUN) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in mmoL/L
Serum creatinine(SCr) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in umoL/L
Urea | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in mmoL/L
Serum alanine transaminase(ALT) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in U/L
Aspartate transaminase(AST) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in U/L
Alkaline phosphatase(ALP) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in U/L
γ-glutamyl transpeptidase (GGT) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in U/L
Total bilirubin(TBIL) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in umoL/L
Total protein(TP) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in g/L
Albumin(ALB) | Day -7(At least 7days before infusion therapy), Day 0 (infusion therapy) , 2 hours after infusion therapy completion
  in g/L

CONTACTS AND LOCATIONS:
Overall Officials: Li ping Liu, Prof., Principal Investigator — Beijing Tiantan Hospital, Captial Medical University
Locations (5):
- China (5):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Sanbo Brain Hospital, Captial Medical University, Beijing, Beijing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality